CLINICAL TRIAL: NCT07356947
Title: The Combined Effect of Mulligan Technique and Scapular Mobilization in Shoulder Adhesive Capsulitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Deraya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Shoulder Adhesive Capsulitis
Record Dates: First submitted 2026-01-13; First posted 2026-01-21 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Adhesive Capsulitis of Shoulder; Frozen Shoulder; Shoulder Pain and Stiffness
Keywords: Adhesive Capsulitis; Frozen Shoulder; Shoulder Joint; Shoulder Pain; Scapulohumeral Rhythm; Mulligan Technique; Mobilization with Movement; Scapular Mobilization
MeSH Terms: conditions — Bursitis; Shoulder Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned into two groups receiving different therapeutic interventions (Mulligan technique with scapular mobilization versus conventional physiotherapy).
Who Masked: Participant
Masking Description: The study is single-blind; participants will not be informed about the treatment group assignment. Groups will be treated and evaluated in separate sessions to maintain blinding.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Physiotherapy (Active Comparator): Participants in this group will receive conventional physiotherapy consisting of:
  Hot pack application for 10 minutes
  Ultrasound therapy in pulsed mode (1 MHz frequency, 0.8 W/cm²) for 5 minutes
  Posterior capsule stretching (2 sets × 3 repetitions, 30-second holds)
  Active and active-assisted range of motion exercises for elevation, internal rotation, external rotation, and pendulum exercises.
  Treatment will be administered three times per week for four weeks. This intervention represents standard physiotherapy care for adhesive capsulitis.
  Interventions: Other: Conventional Physiotherapy
- Mulligan Technique with Scapular Mobilization (Experimental): Participants in this group will receive the Mulligan mobilization technique for shoulder elevation, internal and external rotation, combined with scapular mobilization.
  Each session will include three sets of ten repetitions with a two-minute rest between sets.
  Treatment sessions will occur three times per week for four weeks.
  Interventions: Other: Mulligan Technique with Scapular Mobilization

INTERVENTIONS:
Other: Mulligan Technique with Scapular Mobilization — Participants in this group will receive the Mulligan mobilization technique for shoulder elevation, internal rotation, and external rotation combined with scapular mobilization. Each session will include three sets of ten repetitions with a two-minute rest between sets. Treatment sessions will be conducted three times per week for four weeks. The intervention aims to improve shoulder joint mobility, reduce pain, and enhance scapulohumeral rhythm.
  Arms: Mulligan Technique with Scapular Mobilization
Other: Conventional Physiotherapy — Standard physiotherapy including hot packs, ultrasound, posterior capsule stretching, and active/assisted range-of-motion exercises. Three sessions per week for four weeks.
  Arms: Conventional Physiotherapy

SUMMARY:
The shoulder joint capsule is a fibrous sheath that encloses and stabilizes the structures of the shoulder joint, extending from the anatomical neck of the humerus to the rim of the glenoid fossa. It is normally lax, allowing a wide range of motion. Shoulder adhesive capsulitis, or frozen shoulder, is a common musculoskeletal condition characterized by pain and restricted movement due to thickening and contraction of this capsule. Proper coordination between the scapula and humerus-known as the scapulohumeral rhythm-is essential for normal shoulder motion. Disruption of this rhythm contributes to movement limitation and pain in adhesive capsulitis.

This randomized, single-blind clinical trial aims to investigate the combined effect of the Mulligan technique and scapular mobilization on improving shoulder range of motion, pain, disability, and scapulohumeral rhythm in patients with adhesive capsulitis. Thirty-eight participants aged 30 to 60 years, diagnosed with unilateral adhesive capsulitis, will be randomly assigned to two groups. Group A will receive Mulligan mobilization techniques for shoulder elevation, internal and external rotation, along with scapular mobilization. Group B will receive conventional physical therapy consisting of hot packs, ultrasound, stretching, and range-of-motion exercises. Both groups will undergo treatment three times per week for four weeks.

Primary outcomes include changes in shoulder range of motion (measured using a digital goniometer), pain and disability (measured by the Shoulder Pain and Disability Index [SPADI]), and scapulohumeral rhythm (assessed using tape measurement). The study is expected to provide clinical evidence on whether combining Mulligan and scapular mobilization techniques yields superior functional recovery compared with conventional physiotherapy alone in patients with shoulder adhesive capsulitis.

DETAILED DESCRIPTION:
The shoulder joint capsule is a fibrous structure that surrounds the shoulder joint and connects the anatomical neck of the humerus to the rim of the glenoid fossa. It provides stability to the joint while allowing extensive mobility. In adhesive capsulitis, also known as frozen shoulder, the capsule becomes inflamed, thickened, and contracted, leading to pain, stiffness, and a progressive loss of both active and passive range of motion. This condition is most common in middle-aged individuals and can significantly limit daily function.

Normal shoulder motion depends on a coordinated movement pattern between the scapula and the humerus, known as the scapulohumeral rhythm. During shoulder elevation, approximately two degrees of glenohumeral motion are accompanied by one degree of scapulothoracic movement. Disruption of this rhythm contributes to movement dysfunction, altered biomechanics, and pain. Rehabilitation approaches that restore this coordination are therefore critical for effective management of adhesive capsulitis.

The Mulligan mobilization technique involves the application of sustained accessory glides by the therapist concurrent with the patient's active movement. This technique aims to correct positional faults, reduce pain, and improve joint mobility without provoking discomfort. Scapular mobilization is a manual therapy approach designed to restore normal motion of the scapula on the thoracic cage and to improve the scapulohumeral rhythm during shoulder elevation.

This study is designed as a randomized, single-blind clinical trial to evaluate the combined effect of Mulligan mobilization and scapular mobilization in patients with adhesive capsulitis. Thirty-eight participants aged between 30 and 60 years with unilateral adhesive capsulitis will be randomly assigned into two groups. Group A will receive Mulligan techniques for shoulder elevation, internal rotation, and external rotation in addition to scapular mobilization. Group B will receive conventional physical therapy consisting of hot packs, pulsed ultrasound at 1 MHz and 0.8 W/cm² for five minutes, posterior capsule stretching, and range-of-motion exercises. Both groups will receive therapy three times per week for four weeks.

Outcome assessments will include shoulder range of motion using a digital goniometer, pain and disability using the Shoulder Pain and Disability Index (SPADI), and scapulohumeral rhythm using a tape measurement method. Measurements will be taken before and after the four-week intervention period. It is hypothesized that the combined Mulligan and scapular mobilization protocol will produce greater improvements in pain reduction, joint range, and scapulohumeral coordination compared to conventional physiotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable and willing to provide informed consent to participate in the study.
* Age between 30 and 60 years.
* Both male and female participants.
* Unilateral shoulder involvement with pain and limited active and passive range of motion in lateral rotation, abduction, and internal rotation for more than three months compared with the unaffected side.
* Clinically diagnosed with adhesive capsulitis (frozen shoulder).

Exclusion Criteria:

* History of shoulder surgery.
* History of radiotherapy or chemotherapy.
* Presence of acute infection in the area to be treated.
* History of skin disease.
* History of cervical radiculopathy within the past six months.
* Secondary adhesive capsulitis, rotator cuff tears, shoulder fractures, or dislocations.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in Shoulder Range of Motion (Flexion, Internal Rotation, External Rotation, and Abduction) | Baseline and at 4 weeks post-intervention
  Shoulder joint range of motion (flexion, internal rotation, external rotation, and abduction) will be assessed using a digital goniometer. Each movement will be measured three times, and the mean value will be used for analysis.
Change in Shoulder Pain and Disability (SPADI Score) | Baseline and at 4 weeks post-intervention
  Pain and functional disability will be assessed using the Shoulder Pain and Disability Index (SPADI). The SPADI includes 13 items: a 5-item pain subscale and an 8-item disability subscale. Each item is scored on a 0-10 scale, with higher scores indicating greater pain and disability.
Change in Scapulohumeral Rhythm | Baseline and at 4 weeks post-intervention
  Scapulohumeral rhythm will be evaluated using a tape measurement method during shoulder elevation to assess the coordination between scapular and humeral motion.

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy, Deraya University, Minya, Menia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Norkin C. C., White D. J. Measurement of Joint Motion: A Guide to Goniometry. 5th Edition. F.A. Davis Company; 2016.
- [Background] Kisner C., Colby L. A. Therapeutic Exercise: Foundations and Techniques. 7th Edition. F.A. Davis Company; 2022.
- [Background] Rahbar M, Ranjbar Kiyakalayeh S, Mirzajani R, Eftekharsadat B, Dolatkhah N. Effectiveness of acromioclavicular joint mobilization and physical therapy vs physical therapy alone in patients with frozen shoulder: A randomized clinical trial. Clin Rehabil. 2022 May;36(5):669-682. doi: 10.1177/02692155211070451. Epub 2021 Dec 29. PMID 34964679
- [Background] Brumitt J. Scapula stabilization and rehabilitation exercise prescription. Strength and Conditioning Journal. 2006; 28(3):62-65.
- [Background] McQuade KJ, Smidt GL. Dynamic scapulohumeral rhythm: the effects of external resistance during elevation of the arm in the scapular plane. J Orthop Sports Phys Ther. 1998 Feb;27(2):125-33. doi: 10.2519/jospt.1998.27.2.125. PMID 9475136
- [Background] Mathieu Vanderroost, Venus Pagare, Kai A. Sigel, Naomi O'Reilly, Claire Knott. Scapulohumeral rhythm. Physiopedia. Available online at: https://www.physio-pedia.com/Scapulohumeral_rhythm
- [Background] Ludewig PM, Reynolds JF. The association of scapular kinematics and glenohumeral joint pathologies. J Orthop Sports Phys Ther. 2009 Feb;39(2):90-104. doi: 10.2519/jospt.2009.2808. PMID 19194022
- [Background] Scibek JS, Carcia CR. Assessment of scapulohumeral rhythm for scapular plane shoulder elevation using a modified digital inclinometer. World J Orthop. 2012 Jun 18;3(6):87-94. doi: 10.5312/wjo.v3.i6.87. PMID 22720268
- [Background] Kibler WB. The role of the scapula in athletic shoulder function. Am J Sports Med. 1998 Mar-Apr;26(2):325-37. doi: 10.1177/03635465980260022801. PMID 9548131
- [Background] Sami S. Almureef, et al. Effectiveness of mobilization with conventional physiotherapy in frozen shoulder patients: a systematic review. Journal of Musculoskeletal Research. 2020.